CLINICAL TRIAL: NCT07334028
Title: Observational Study to Ascertain the Optimum Time to Observe the Infra-red Image of Varicose Veins in the Lower Limb When Standing From a Supine Position.
Brief Title: Study to Find Out the Timing for the Optimal Imaging of Varicose Veins Using Infrared Thermography.
Status: Recruiting | Type: Observational
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Principal Investigator, Mark Whiteley, Consultant Venous Surgeon, The Whiteley Clinic
Other Study IDs: TWC-IR-TAGSS-001
Record Dates: First submitted 2025-09-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Varicose Veins Leg
Keywords: varicose vein; infrared imaging
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients presenting with varicose veins: Primary or recurrent varicose veins
  Interventions: Diagnostic Test: Infrared imaging

INTERVENTIONS:
Diagnostic Test: Infrared imaging — Patients will only have infrared images taken of their legs

SUMMARY:
The goal of this observational study is to identify the optimal time of Infrared imaging of varicose veins when patients move from a lying to a standing position.

The primary purpose is to enable us to improve our imaging of varicose veins in patients presenting with primary or recurrent leg varicose veins.

The main questions it aims to answer are:

Outcome measure 1- How long after standing up from lying supine do leg varicose veins show up best on infrared imaging? Outcome measure 2 - Is there any difference in this timing between varicose veins arising from different sources in the leg?

Patients will be asked to stand, and sequential infrared images will be taken every 5 seconds for 3 minutes.

DETAILED DESCRIPTION:
Patients who are having a Duplex ultrasound of their lower-limb veins for the assessment of varicose veins (primary or recurrent) and who have consented to participation in the study will be taken from the scanning room to the research room (within 20 meters).

The patient will be asked for their height and weight to enable BMI to be calculated. The patient will then lie down horizontally for 5 minutes on a bed in the research room. At the end of the 5 minutes, an IR image will be taken of the participant's lower limbs to ensure clearance of varicose veins.

The patient will then be asked to stand in front of an IR camera on a mat with marked positions for their feet on the floor in a position ensuring maximum surface area coverage of lower-limb varicose veins by the camera. The patient will stand still for a period of 3 minutes whilst the IR camera (HIKMICRO M10) takes a series of JPEG photos every 5 seconds. The position of the camera will be adjusted so that the top of the image is at the level of the hip, and the bottom of the image at the sole of the foot. Hence, the image size will be maximised to include the whole leg.

The first image will be taken immediately the patient stands and is in position, minimising any lag and aiming to be within 5 seconds of starting to move from the supine position. After 3 minutes, the patient will be able to sit down and then return to the consultation room.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing venous duplex ultrasound scan for suspected varicose veins (primary or recurrent).
* Able to stand still for 5 minutes.
* Able to get on to and off of the surgical couch unaided.
* Patient giving consent.

Exclusion Criteria:

* Refusing consent.
* Unable to get on a couch or stand unaided.
* Unable to stand still for 5 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient attending our vein clinc for assessement of their varicose veins
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Time of optimal Infrared imaging of leg varicose veins after standing from lying | The whole process for the patient will be a maximum of 20 minutes. The analysis of all of the images will be completed within 1 month of the end of the data collection.
  Sequential infrared images will show us at what time point the optimal infrared images have been obtained.

SECONDARY OUTCOMES:
Variation of optimal infrared image timing due to the source of venous reflux | The patient data collection will be within 20 minutes, and the analysis within 1 month.
  Using the infrared images and comparing them with the duplex ultrasound scans that the patient is having as part of their normal medical assessment, we will subdivide the images by the underlying source of the varicose veins and venous reflux. We will assess whether there is a different time to optimal Infrared imaging with different patterns of venous reflux, predominantly great or small saphenous reflux.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS FRCS(Gen) MBBS, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD is not relevant to the outcomes

REFERENCES:
- [Background] Brian Meneses-Claudio, W. A.-D.-G. (2019). Detection of Suspicions of Varicose Veins in the Legs using Thermal Imaging. International Journal of Advanced Computer Science and Applications(IJACSA). doi:10.14569/IJACSA.2019.0100554